CLINICAL TRIAL: NCT06286540
Title: Efficacy and Safety of Lymphoblock in the Prevention of Postoperative Lymphorrhea After Surgical Treatment of the Thoracoabdominal Aorta: a Single-center, Randomized, Placebo-controlled, Double-blind Study.
Brief Title: Evaluation of the Efficacy and Safety of Surgical Device "Lymphoblock" for Prevention of Lymphorrhea in Patients With Thoracoabdominal Aorta Repair.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Petrovsky National Research Centre of Surgery (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 26031993
Record Dates: First submitted 2024-02-22; First posted 2024-02-29 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Aorta Abdominalis; Aneurysm; Aorta Thoracic; Aneurysm
MeSH Terms: conditions — Aortic Aneurysm, Abdominal; Aortic Aneurysm, Thoracic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lymphoblock (Experimental): Patients from this group received Lymphoblock.
  Interventions: Device: Lymphoblock
- Placebo (Placebo Comparator): Patients from this group received placebo.
  Interventions: Device: Placebo

INTERVENTIONS:
Device: Lymphoblock — 1 time per surgery with the exposition for 20 minutes.
  Arms: Lymphoblock
Device: Placebo — 1 time per surgery with the exposition for 20 minutes.
  Arms: Placebo

SUMMARY:
Randomized, double-blind, placebo-controlled study will determine the clinical efficacy and safety of Lymphoblock in the prevention of postoperative retroperitoneal chylo-/lymphorrhoea in patients with open surgical treatment of the thoracoabdominal aorta. It is planned to recruit 138 clinical observations. Efficacy will be evaluated based on clinical and laboratory data.

DETAILED DESCRIPTION:
The study design will include patients with open surgical repair of the thoracoabdominal aorta who underwent thoracophrenolumbotomy with retroperitoneal exposure of the aorta. It is assumed the lymphoblock to reduce the incidence of postoperative lympho-/chylorrhea. Patients will be divided based on randomization into groups that will receive a lymphoblock or a placebo. It is planned to recruit 138 patients, 69 patients in each group. The drug will be used right before wound closure. The solution will be applied to the surface of the wound with further exposure and draining. Blood test and drainage discharge parameters (from the left pleural cavity and retroperitoneum) will be examined in postoperative period. The thoracic and abdominal CT and ultrasound will be performed to exclude presence of effusion and/or lymphocele.

ELIGIBILITY:
Inclusion Criteria:

* patient in thoracoabdominal or abdominal aorta repair underwent retroperitoneal aortic access

Exclusion Criteria:

* refusal to participate in the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Estimated)
Dates: Start 2023-02-22 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Chylous Effusion (Сhilo-/lymphorrhea) | within 10 days of starting a regular diet after surgery
  This outcome will be determined by assessing the milky of the drainage discharge, and comparing the content of triglycerides, glucose, cholesterol and lactate dehydrogenase (LDH) in the drainage discharge with those in the blood plasma
Number of Participants with Lymphocele | 10 days after the surgery in patient who starting a regular diet after drainage removal
  retroperitoneal liquid formation ≥5 cm in diameter according to ultrasound after drainage removal

SECONDARY OUTCOMES:
The amount of drainage discharge 1 | 24 hours after the surgery
  volume of drainage discharge obtained in the first 24 hours after surgery, measured in milliliters (ml)
The amount of drainage discharge 2 | 48 hours after the surgery
  volume of drainage discharge obtained in the first 48 hours after surgery, measured in milliliters (ml)
The amount of drainage discharge 3 | 72 hours after the surgery
  volume of drainage discharge obtained in the first 72 hours after surgery, (ml)
Concentration of triglycerides in the drainage discharge | 72 hours after the surgery
  count of triglycerides in the drainage discharge, received from drainage tube, (mg/dL)
Concentration of triglycerides in blood plasma | 72 hours after the surgery
  count of triglycerides in the blood plasma, (mg/dL)
Concentration of cholesterol in the drainage discharge | 72 hours after the surgery
  count of cholesterol in the drainage discharge, received from drainage tube, (mg/dL)
Concentration of cholesterol in the blood plasma | 72 hours after the surgery
  count of cholesterol in the blood plasma, (mg/dL)
Concentration of protein in the drainage discharge | 72 hours after the surgery
  count of total protein in the drainage discharge, received from drainage tube, (g/dL)
Concentration of protein in the blood plasma | 72 hours after the surgery
  count of total protein in the blood plasma, (g/dL)
Concentration of albumin in the drainage discharge | 72 hours after the surgery
  count of albumin in the drainage discharge, received from drainage tube, (g/dL)
Concentration of albumin in the blood plasma | 72 hours after the surgery
  count of albumin in the blood plasma, (g/dL)
Concentration of lactate dehydrogenase in the drainage discharge | 72 hours after the surgery
  count of albumin in the drainage discharge, received from drainage tube (IU/L)
Concentration of lactate dehydrogenase in the blood plasma | 72 hours after the surgery
  count of lactate dehydrogenase in the blood plasma (IU/L)
Concentration of glucose in the drainage discharge | 72 hours after the surgery
  Content of glucose in the drainage discharge, received from drainage tube, (mg/dL)
Concentration of glucose in the blood plasma | 72 hours after the surgery
  Content of glucose in the blood plasma (mg/dL)
Number of Participants with Pleural effusion within 10 days | 10 days after the surgery in patient who starting a regular diet after drainage removal
  left pleural fluid accumulations (≥500 ml) after drainage removal drainage removal
Number of Participants with Lymphocele 3 months after the surgery | 3 months after the surgery
  liquid formation ≥5 cm in diameter according to ultrasound after drainage removal
Number of Participants with Pleural effusion 3 months after the surgery | 3 months after the surgery
  left pleural fluid accumulations (≥500 ml) after drainage removal

CONTACTS AND LOCATIONS:
Overall Officials: Eduard Charchyan, MD, Principal Investigator — Petrovsky NRCS
Locations (1):
- Petrovsky NRCS, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No